CLINICAL TRIAL: NCT06196034
Title: Genetic Association With Various Severities, Phenotypes and Endotypes of Asthma.
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Dr, Chinese University of Hong Kong
Other Study IDs: Asthma Genetics_V2_08Aug2023
Record Dates: First submitted 2023-12-23; First posted 2024-01-09 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for genetics study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma: Subjects with asthma
  Interventions: Genetic: No intervention
- Control: Subjects with no asthma
  Interventions: Genetic: No intervention

INTERVENTIONS:
Genetic: No intervention — No intervention

SUMMARY:
There is limited information on genetics associated with asthma in Chinese. An earlier meta-analysis found that ADAM33, FcεRIb, RANTES, TNF-a, ACE, b2-AR, IL-4R and IL-13 genes could be proposed as asthma susceptible genes in the Chinese population. However, given the limited number of studies, more data are required to validate these associations.

Future research must address key issues such as the broad clinical variability of asthma and the underrepresentation of populations of non-European heritage. Endotype-specific SNPs and unique biological insights may be obtained by conducting GWAS/EWAS on homogeneous populations of more therapy-resistant T2-low, adult-onset, obesity-associated asthma or asthma with particular co-morbidities.

The primary objective is to investigate the association between genetic polymorphisms and various severities of asthma.

DETAILED DESCRIPTION:
Currently, many studies on asthma genetics are limited by the dominance of populations of European descent. In addition, there are few genetic studies that focus on moderate-to-severe asthma.

There is limited information on genetics associated with asthma in Chinese. An earlier meta-analysis found that ADAM33, FcεRIb, RANTES, TNF-a, ACE, b2-AR, IL-4R and IL-13 genes could be proposed as asthma susceptible genes in the Chinese population. However, given the limited number of studies, more data are required to validate these associations.

Future research must address key issues such as the broad clinical variability of asthma and the underrepresentation of populations of non-European heritage. Endotype-specific SNPs and unique biological insights may be obtained by conducting GWAS/EWAS on homogeneous populations of more therapy-resistant T2-low, adult-onset, obesity-associated asthma or asthma with particular co-morbidities.

Objectives Primary objective To investigate the association between genetic polymorphisms and various severities of asthma (e.g. mild, moderate, severe).

Secondary objectives

1. Identify the most common genetic variants associated with asthma in Chinese patients.
2. Determine the frequency and distribution of these genetic variants in Chinese patients compared to healthy controls.
3. Explore the potential interactions between genetic and environmental factors in the development of asthma in Chinese patients.
4. Explore the frequency and distribution of these genetic variants in patients with various phenotypes and endotypes (examples: including TH2 high asthma, Asthma COPD overlap, poor lung function, onset of illness)

This is a prospective observational study in outpatients with asthma seen and treated by physicians in the Prince of Wales Hospital. A total of 1000 asthma patients will be enrolled, along with 1000 controls matched for age, sex, and ethnicity. All participants will provide blood samples for genetic analysis, and clinical data will be collected from medical records and patient interviews. Genetic variants will be genotyped using high-throughput sequencing methods.

ELIGIBILITY:
Inclusion Criteria:

* • All patients with confirmed diagnosis of asthma (defined as those with a consistent history and prior documented evidence of variable airflow obstruction, with evidence of an increase in FEV1 greater than 12% or 400 mL following bronchodilator or bronchial hyperresponsiveness on bronchial provocation testing, when stable) 12

  * Able to sign written informed consent form to participate in the study.

Exclusion Criteria:

* • Patients currently with acute exacerbation of asthma by GINA guideline. (For subjects with asthma exacerbation, they can join the study after 6 weeks post recovery from the exacerbation.)

  * Patients with respiratory diseases that can show similar symptoms to chronic airway diseases such as bronchiectasis, tuberculosis(TB)-destroyed lung parenchyma, endobronchial TB, and lung cancer, or those who have history of these diseases based on physician's judgment.
  * Patients currently diagnosed with pneumonia and acute bronchitis.

For control subject: the inclusion will be having no clinical diagnosis of asthma.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study in outpatients with asthma seen and treated by physicians in the Prince of Wales Hospital. A total of 1000 asthma patients will be enrolled, along with 1000 controls matched for age, sex, and ethnicity.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-01-04 (Estimated); Study Completion 2029-01-04 (Estimated)

PRIMARY OUTCOMES:
association between genetic polymorphisms and various severities of asthma | 3 years
  association between genetic polymorphisms and various severities of asthma

SECONDARY OUTCOMES:
Identify the most common genetic variants associated with asthma in Chinese patients. | 3 years
  Identify the most common genetic variants associated with asthma in Chinese patients.
Explore the frequency and distribution of these genetic variants in patients with various phenotypes and endotypes | 3 years
  Explore the frequency and distribution of these genetic variants in patients with various phenotypes and endotypes (examples: including TH2 high asthma, Asthma COPD overlap, poor lung function, onset of illness)

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, Study Director — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - The Chinese University of Hong Kong, Hong Kong, New Territories
  - The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
We can share the data (no patient identity reviewed) if there are projects (with reasonable quality and request) requesting that according to the rules of our institution.